CLINICAL TRIAL: NCT03590808
Title: Efficacy and Safety of Influenza Vaccine in Cancer Patients Receiving Immune Checkpoint Inhibitor
Brief Title: Influenza Vaccination in Patients Receiving Immune Checkpoint Inhibitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: Principal Investigator, Wan Beom Park, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1806-088-951
Record Dates: First submitted 2018-07-10; First posted 2018-07-18 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Influenza; Solid Carcinoma
Keywords: Influenza; vaccine; solid carcinoma; immune checkpoint; efficacy; safety
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Double center prospective case-control clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immune checkpoint inhibitor (Experimental): Solid cancer patients who receiving immune checkpoint inhibitor patients
  will be undergone "Influenza vaccination" using purified inactivated influenza virus antigen (Green Cross Corp.) 0.5 mL IM once
  Interventions: Biological: Influenza vaccination
- Cytotoxic chemotherapy (Active Comparator): Solid cancer patients who receiving conventional cytotoxic chemotherapy
  will be undergone "Influenza vaccination" using purified inactivated influenza virus antigen (Green Cross Corp.) 0.5 mL IM once
  Interventions: Biological: Influenza vaccination

INTERVENTIONS:
Biological: Influenza vaccination — Purified inactivated influenza virus antigen (Green Cross Corp) 0.5 mL once IM

SUMMARY:
The purpose of this study is to elucidate efficacy and safety of influenza vaccine in cancer patients receiving immune checkpoint inhibitor.

DETAILED DESCRIPTION:
* Solid cancer patients receiving immune checkpoint inhibitor or cytotoxic chemotherapy will be recruited 1:2 manner in two hospitals. Target numbers are 48 and 95, respectively.
* All the participants will be vaccinated for influenza during their chemotherapy when they meet inclusion criteria.
* All the participants will be asked if they have any contraindication for influenza vaccine by a physician before vaccination.
* Hemagglutination inhibition Ab titre at pre-vaccination and post-vaccination (21-35 days after vaccination) will be examined in all participants to examine seroprotection rates, seroconversion rates, and changes in geometric mean titer.
* And they will be monitored for any vaccination-related adverse reaction or immune-related adverse events after 2-4 days(via phone call), and till 6 months after vaccination (when they visit oncology clinics).

ELIGIBILITY:
Inclusion Criteria:

* Solid cancer patients receiving immune checkpoint inhibitor or cytotoxic chemotherapeutic agent in Seoul National University Hospital or Seoul National University Bundang Hospital.
* Patients who was not vaccinated for influenza in 2018-2019 season
* ECOG performance status 0 or 1
* Patients who fulfilling following laboratory criteria Total bilirubin ≤ 1.5 x upper normal limit Aspartate transaminase, alanine transaminase ≤ 2.5 x upper normal limit Alkaline phosphatase ≤ 2.5 x upper normal limit Creatinine ≤ upper normal limit
* Patients who can understand and agreed with the informed consents.

Exclusion Criteria:

* Patients having contraindication for influenza vaccination (e.g. egg allergy)
* Patients who receive any immunosuppressant (excluding steroid for anti-emetic effect)
* Patients with HIV infection
* Patients with autoimmune disease who are anticipated to have a problem with immunogenicity for vaccine
* Patients who have transplanted organ and receive immunosuppressants
* Patients who are suspected to have active infection (e.g. pneumonia)
* Patients who receive targeted chemotherapeutic agent alone for cancer treatment
* Patients who could not receive cancer chemotherapy due to hematologic abnormality at the date of the participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate | 21 to 35 days after vaccination
  The percentage of vaccine recipients with a serum haemagglutination inhibition(HI) titre ≥40 post vaccination (21-28 days)

SECONDARY OUTCOMES:
Seroconversion rate | 21 to 35 days after vaccination
  Seroconversion rate is defined as the percentage of vaccine recipients with a fourfold increase or more in post-vaccination HI titre
Geometric mean titer of HI | 21 to 35 days after vaccination
  Geometric mean titers of HI (haemagglutination inhibition) after vaccination
Injection-related adverse events | 21 to 35 days after vaccination
  The proportion of patients who experienced local or systemic adverse events related to vaccination
Immune-related adverse events | 6 months after vaccination
  The proportion of patients who experienced immune checkpoint inhibitor induced immune-related adverse events
T-cell mediated immune response | 21 to 35 days after vaccination
  The levels of intracellular cytokines measured by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Wan Beom Park, M.D., PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
We are not planning to share IPDs publically, but de-identified individual participant data for all outcome measures could be shared with other researchers under their request.

REFERENCES:
- [Background] Postow MA, Sidlow R, Hellmann MD. Immune-Related Adverse Events Associated with Immune Checkpoint Blockade. N Engl J Med. 2018 Jan 11;378(2):158-168. doi: 10.1056/NEJMra1703481. No abstract available. PMID 29320654
- [Background] Adelstein D, Gillison ML, Pfister DG, Spencer S, Adkins D, Brizel DM, Burtness B, Busse PM, Caudell JJ, Cmelak AJ, Colevas AD, Eisele DW, Fenton M, Foote RL, Gilbert J, Haddad RI, Hicks WL, Hitchcock YJ, Jimeno A, Leizman D, Lydiatt WM, Maghami E, Mell LK, Mittal BB, Pinto HA, Ridge JA, Rocco J, Rodriguez CP, Shah JP, Weber RS, Witek M, Worden F, Yom SS, Zhen W, Burns JL, Darlow SD. NCCN Guidelines Insights: Head and Neck Cancers, Version 2.2017. J Natl Compr Canc Netw. 2017 Jun;15(6):761-770. doi: 10.6004/jnccn.2017.0101. PMID 28596256
- [Background] Ettinger DS, Wood DE, Aisner DL, Akerley W, Bauman J, Chirieac LR, D'Amico TA, DeCamp MM, Dilling TJ, Dobelbower M, Doebele RC, Govindan R, Gubens MA, Hennon M, Horn L, Komaki R, Lackner RP, Lanuti M, Leal TA, Leisch LJ, Lilenbaum R, Lin J, Loo BW Jr, Martins R, Otterson GA, Reckamp K, Riely GJ, Schild SE, Shapiro TA, Stevenson J, Swanson SJ, Tauer K, Yang SC, Gregory K, Hughes M. Non-Small Cell Lung Cancer, Version 5.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Apr;15(4):504-535. doi: 10.6004/jnccn.2017.0050. PMID 28404761
- [Background] Motzer RJ, Jonasch E, Agarwal N, Bhayani S, Bro WP, Chang SS, Choueiri TK, Costello BA, Derweesh IH, Fishman M, Gallagher TH, Gore JL, Hancock SL, Harrison MR, Kim W, Kyriakopoulos C, LaGrange C, Lam ET, Lau C, Michaelson MD, Olencki T, Pierorazio PM, Plimack ER, Redman BG, Shuch B, Somer B, Sonpavde G, Sosman J, Dwyer M, Kumar R. Kidney Cancer, Version 2.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Jun;15(6):804-834. doi: 10.6004/jnccn.2017.0100. PMID 28596261
- [Background] Keam B, Kim MK, Choi Y, Choi SJ, Choe PG, Lee KH, Kim TM, Kim TY, Oh DY, Kim DW, Im SA, Kim NJ, Heo DS, Park WB, Oh MD. Optimal timing of influenza vaccination during 3-week cytotoxic chemotherapy cycles. Cancer. 2017 Mar 1;123(5):841-848. doi: 10.1002/cncr.30468. Epub 2016 Dec 20. PMID 27997703
- [Background] Fiore AE, Uyeki TM, Broder K, Finelli L, Euler GL, Singleton JA, Iskander JK, Wortley PM, Shay DK, Bresee JS, Cox NJ; Centers for Disease Control and Prevention (CDC). Prevention and control of influenza with vaccines: recommendations of the Advisory Committee on Immunization Practices (ACIP), 2010. MMWR Recomm Rep. 2010 Aug 6;59(RR-8):1-62. PMID 20689501
- [Background] Pollyea DA, Brown JM, Horning SJ. Utility of influenza vaccination for oncology patients. J Clin Oncol. 2010 May 10;28(14):2481-90. doi: 10.1200/JCO.2009.26.6908. Epub 2010 Apr 12. PMID 20385981
- [Background] Dueck AC, Mendoza TR, Mitchell SA, Reeve BB, Castro KM, Rogak LJ, Atkinson TM, Bennett AV, Denicoff AM, O'Mara AM, Li Y, Clauser SB, Bryant DM, Bearden JD 3rd, Gillis TA, Harness JK, Siegel RD, Paul DB, Cleeland CS, Schrag D, Sloan JA, Abernethy AP, Bruner DW, Minasian LM, Basch E; National Cancer Institute PRO-CTCAE Study Group. Validity and Reliability of the US National Cancer Institute's Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). JAMA Oncol. 2015 Nov;1(8):1051-9. doi: 10.1001/jamaoncol.2015.2639. PMID 26270597
- [Derived] Keam B, Kang CK, Jun KI, Moon SM, Suh KJ, Lee DW, Ock CY, Kim M, Choi Y, Lim Y, Lee KH, Kim SH, Kim TM, Kim TY, Oh DY, Kim DW, Im SA, Lee JS, Kim ES, Kim HB, Kim NJ, Kim YJ, Park WB, Oh MD. Immunogenicity of Influenza Vaccination in Patients with Cancer Receiving Immune Checkpoint Inhibitors. Clin Infect Dis. 2020 Jul 11;71(2):422-425. doi: 10.1093/cid/ciz1092. PMID 31680143